CLINICAL TRIAL: NCT01201395
Title: Longitudinal Study of Repaired or Replaced Dental Restorations
Brief Title: DPBRN Longitudinal Study of Repaired or Replaced Dental Restorations
Status: Completed | Type: Observational
Sponsor: Dental Practice-Based Research Network (Network)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); HealthPartners Institute (Other); Kaiser Permanente (Other); Permanente Dental Associates Group, Oregon (Other); University of Alabama at Birmingham (Other); University of Florida (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Gregg H. Gilbert, DDS, MBA, FAAHD, Professor and Chair, Department of General Dental Sciences, Dental Practice-Based Research Network
Other Study IDs: 111010; U01DE016747 (NIH)
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Dental Caries
Keywords: Dental Caries; Assessment; dental materials
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dental caries assessment

SUMMARY:
The purpose of this study is to assess the quality and expected lifespan of fillings recorded in the DPBRN "Reasons for replacement and repair of dental restorations" study, and the factors affecting how long the fillings last.

DETAILED DESCRIPTION:
The study is an observational follow-up of previously placed dental restorations (fillings)and is conducted during routing dental care visits.

ELIGIBILITY:
Inclusion Criteria:

* participant in the DPBRN "Reasons for replacement or repair of dental restorations" study

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The participants directly involved in this study are the particpants who have sought dental treatment in the practitioner-investigators' practices and participated in the DPBRN "Reasons for replacement or repair of dental restorations" study.
Sampling Method: Non-Probability Sample
Enrollment: 9813 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valeria V Gordan, DDS, MS, Principal Investigator — University of Florida
Locations (7):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida College of Dentistry, Gainesville, Florida
  - Health Partners Dental Group, Minneapolis, Minnesota
  - Health Partners Research Foundation, Minneapolis, Minnesota
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Permanente Denrtal Associates, Portland, Oregon
- University of Copenhagen Royal Dental College, Copenhagen, Denmark

REFERENCES:
- See also: Dental Practice-Based Research Network — http://DPBRN.org
- See also: Dental Practice-Based Research Network — http://DentalPBRN.org